CLINICAL TRIAL: NCT04343339
Title: Evolution of Psychoactive Substances Consumption in Connection With COVID-19 Containment - EPILOGUE
Brief Title: Evolution of Psychoactive Substances Consumption in Connection With COVID-19 Containment
Acronym: EPILOGUE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0195
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-04

CONDITIONS: Addiction, Substance; COVID-19
Keywords: Risk of overdose on de-confinment; COVID-19 containment will change drugs practices; COVID-19 containment will changes access to care; Addiction is a common disease; Alcohol; Containment; Drug use
MeSH Terms: conditions — Substance-Related Disorders; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current containment linked to COVID-19 will have consequences for people suffering from addiction and there is a risk of overdoses when the containment ends. So the investigators hypothesize that this health crisis is an opportunity to develop risk reduction and access to care for vulnerable people who lives with an addiction.

The main objective of this study is to describe the changes in the psychoactive substances consumption during the containment in people suffering from addiction. The secondary objectives are to describe the evolution at 1 month from the end of the containment of problematic consumption and the level of access to care of these users

ELIGIBILITY:
Inclusion criteria:

* >18 years
* Accept study
* live with an addiction

Exclusion criteria:

- not being able to answer the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Person who lives with an addiction accepting the principle of the study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Evolution of consumption | 1 day
  measurement of the difference in drugs consumption caused by containment (delta)
Evolution of consumption | 1 month after confinmant
  measurement of the difference in drugs consumption caused by containment (delta)

SECONDARY OUTCOMES:
health care access | 1 day
  number of drug users referred to care (%)
health care access | 1 month after confinmant
  number of drug users referred to care (%)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Donnadieu-Rigole, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC